CLINICAL TRIAL: NCT02357004
Title: Mechanisms of Refractory Hypertension (Carvedilol)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in priority of interventional protocols
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, David Calhoun, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A000502641
Record Dates: First submitted 2015-01-22; First posted 2015-02-06 (Estimated); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Hypertensive
MeSH Terms: interventions — Carvedilol; Chlorthalidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carvedilol (Experimental): Carvedilol CR 40 mg daily in addition to their normal BP medications. Subjects will be seen in follow-up at 2-week intervals for the duration of the 8-week intervention period. If the clinic BP remains elevated (>140/90 mmHg) at any of the follow-up visits, the study medication will be titrated up to carvedilol CR 80 mg daily (subjects will take 2 of the study pills).
  Interventions: Drug: Carvedilol
- Chlorthalidone (Experimental): Chlorthalidone 12.5 mg daily in addition to their normal BP medications. Subjects will be seen in follow-up at 2-week intervals for the duration of the 8-week intervention period. If the clinic BP remains elevated (>140/90 mmHg) at any of the follow-up visits, the study medication will be titrated up to chlorthalidone 25 mg daily (subjects will take 2 of the study pills).
  Interventions: Drug: Chlorthalidone

INTERVENTIONS:
Drug: Carvedilol — CR 40 mg daily in addition to normal BP medications
  Arms: Carvedilol
Drug: Chlorthalidone — 12.5 mg daily in addition to normal BP medications
  Arms: Chlorthalidone

SUMMARY:
The purpose of this protocol is test whether patients with hypertension refractory to antihypertensive treatment have evidence of excessive sympathetic (i.e., nervous system) activity.

DETAILED DESCRIPTION:
Refractory hypertension refers to high blood pressure that is failing conventional antihypertensive therapies. In a retrospective assessment of such patients in our clinic we observed that resting clinic heart rates were higher in patients with refractory hypertension compared to patients with controlled hypertension. This observation has led to the hypothesis that refractory hypertension is caused by excessive sympathetic output. This protocol is designed to test this hypothesis by comparing the BP response to carvedilol verses chlorthalidone in patients with refractory hypertension. If their extreme treatment resistance is neurogenic is etiology, a significantly larger BP response to carvedilol should occur compared to chlorthalidone.

ELIGIBILITY:
Inclusion Criteria:

* Uncontrolled clinic BP (>140/90 mmHg)
* Receiving 5 or more antihypertensive agents including an ACE inhibitor or ARB, calcium channel blocker, and chlorthalidone 25 mg

Exclusion Criteria:

* Current use of an alpha or beta or combined alpha-beta antagonist
* Known allergy to alpha-beta antagonists
* CKD (eGFR <40 ml/min/m2)
* MI, stroke or episode of CHF exacerbation within 3 months
* Bradycardia <50 bpm; history of 2nd or 3rd degree heart block unless treated by a pacemaker
* Pregnant or breast-feeding women
* Known hypersensitivity to chlorthalidone or other sulfonamide-derived drugs

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
% of subjects who achieve BP control (<140/90 mm Hg) | 8 weeks after baseline
  BP will be measured 8 weeks after starting carvedilol and after starting chlorthaidone. The percent of subjects with BP of <140/90 mm HG in each group will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: David A. Calhoun, MD, Principal Investigator — Cardiology Department - University of Alabama at Birmingham